CLINICAL TRIAL: NCT00856206
Title: A Multi-Center, Randomized, Double-Blind, Placebo Controlled Trial of the Safety of Rilonacept for the Prophylaxis of Gout Flares in Patients on Urate- Lowering Therapy
Brief Title: Review of Safety Using Rilonacept in Preventing Gout Exacerbations (RE-SURGE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IL1T-GA-0815
Record Dates: First submitted 2009-02-21; First posted 2009-03-05 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Gout
Keywords: Metabolism, Inborn Errors; Allopurinol; Metabolic Disease; Genetic Diseases, Inborn; Musculoskeletal Diseases; Joint Diseases; Arthritis; Rheumatic Diseases; Metabolic disorder; Purine Pyrimidine Metabolism, Inborn Errors; Gout; Intercritical Gout
MeSH Terms: conditions — Gout; Metabolism, Inborn Errors; Metabolic Diseases; Genetic Diseases, Inborn; Musculoskeletal Diseases; Joint Diseases; Arthritis; Rheumatic Diseases; Purine-Pyrimidine Metabolism, Inborn Errors | interventions — rilonacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Two subcutaneous injections of Placebo (for Rilonacept) as a loading dose on Day 1 followed by a single injection once a week (qw) from Week 1 to Week 15.
  Interventions: Other: Placebo
- Rilonacept 160 mg (Experimental): Two subcutaneous injections of Rilonacept 160 mg (for a total of 320 mg) as a loading dose on Day 1, followed by a single 160 mg injection of Rilonacept qw from Week 1 to Week 15.
  Interventions: Biological: Rilonacept

INTERVENTIONS:
Biological: Rilonacept — Rilonacept 160 mg subcutaneous injection once a week
  Arms: Rilonacept 160 mg
Other: Placebo — Placebo subcutaneous injection once a week
  Arms: Placebo

SUMMARY:
The purpose of this clinical research study is to determine the safety and effectiveness of an experimental drug called rilonacept in subjects with gout who are on urate-lowering therapy. Subjects will participate in this study for approximately 20 weeks. Rilonacept is being studied for use in preventing gout flares in subjects on urate-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 80 years of age;
* Previously met the preliminary criteria of American Rheumatism Associatio (ARA) for the classification of acute gout arthritis of primary gout;
* Subjects with history of gout, initiating or currently on urate lowering; therapy who are at risk of gout flare.

Exclusion Criteria:

* Acute gout flare within 2 weeks prior to the screening visit and during the screening visit;
* Persistent chronic or active infections;
* History of an allergic reaction to allopurinol;
* History or presence of cancer within 5 years of the Screening Visit;;;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1315 (Actual)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Evans, PharmD, Study Director — Regeneron Pharmaceuticals
Locations (124):
- United States (77):
  - Alabaster, Alabama
  - Mesa, Arizona
  - Burbank, California
  - Long Beach, California
  - Los Angeles, California
  - Upland, California
  - Brooksville, Florida
  - Clearwater, Florida
  - DeBary, Florida
  - DeLand, Florida
  - Jacksonville, Florida
  - Naples, Florida
  - Palm Harbor, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Canton, Georgia
  - Decatur, Georgia
  - Sandy Springs, Georgia
  - Stockbridge, Georgia
  - Boise, Idaho
  - Brownsburg, Indiana
  - Evansville, Indiana
  - Greenfield, Indiana
  - Bowling Green, Kentucky
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Springfield, Massachusetts
  - Worcester, Massachusetts
  - Bingham Farms, Michigan
  - Brooklyn Center, Minnesota
  - Richmond Heights, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Kalispell, Montana
  - Lincoln, Nebraska
  - Elizabeth, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Mineola, New York
  - New York, New York
  - Roslyn, New York
  - Durham, North Carolina
  - Hickory, North Carolina
  - Mooresville, North Carolina
  - Morganton, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Middleburg Heights, Ohio
  - Duncansville, Pennsylvania
  - Morrisville, Pennsylvania
  - Ridley Park, Pennsylvania
  - Willow Grove, Pennsylvania
  - Anderson, South Carolina
  - Monck's Corner, South Carolina
  - Orangeburg, South Carolina
  - Johnson City, Tennessee
  - Arlington, Texas
  - Carrollton, Texas
  - Corsicana, Texas
  - Dallas, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - San Antonio, Texas
  - Southlake, Texas
  - Sugarland, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Oak Creek, Wisconsin
  - Wauwatosa, Wisconsin
- Germany (7):
  - Künzing, Bavaria
  - Hamburg, Hamburg
  - Dietzenbach, Hesse
  - Essen, North Rhine-Westphalia
  - Goch, North Rhine-Westphalia
  - Siegen, North Rhine-Westphalia
  - Rhaunen, Rhineland-Palatinate
- India (8):
  - Secundrabad, Andh Prad
  - Ahmedabad, Gujarat
  - Gandhinagar, Gujarat
  - Bangalore, Karna
  - Mangalore, Karna
  - Mumbai, Mahara
  - New Dehli, National Capital Territory of Delhi
  - Kolkata, West Bengal
- Indonesia (7):
  - Denpasar, Bali
  - Makassar, South Sulawesi
  - Padang, West Sumatra
  - Bandung
  - Malang
  - South Sumatra
  - Yogyakarta
- South Africa (21):
  - Port Elizabeth, E Cape
  - Bloemfontein, Free State
  - Benoni, Gauteng
  - Centurion, Gauteng
  - Eldoraigne, Gauteng
  - Johannesburg, Gauteng
  - Kempton Park, Gauteng
  - Krugersdorp, Gauteng
  - Lenasia, Gauteng
  - Limpopo, Gauteng
  - Pretoria, Gauteng
  - Rustenburg, Gauteng
  - Soweto, Gauteng
  - Dundee, KZ-Natal
  - Durban North, KZ-Natal
  - Phoenix, KZ-Natal
  - Verulam, KZ-Natal
  - Breyten, Mpumalanga
  - Durban, Mpumalanga
  - Cape Town, W Cape
  - Mpumalanga
- Taiwan (4):
  - Changhua
  - Hualien City
  - Tainan
  - Taipei

REFERENCES:
- [Derived] Sundy JS, Schumacher HR, Kivitz A, Weinstein SP, Wu R, King-Davis S, Evans RR. Rilonacept for gout flare prevention in patients receiving uric acid-lowering therapy: results of RESURGE, a phase III, international safety study. J Rheumatol. 2014 Aug;41(8):1703-11. doi: 10.3899/jrheum.131226. Epub 2014 Jul 15. PMID 25028379

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 71 study sites in United States and rest of world (ROW) between 23 March 2009 and 14 January 2011. A total of 2311 participants were screened in the study.
Pre-assignment Details: Out of 2311 participants, 1315 were randomized and treated in the study. Participants were randomized in 3:1 ratio to receive Rilonacept 160 mg or placebo.
Period: Overall Study
Arm/Group | Placebo | Rilonacept 160 mg
Started | 330 | 985
Completed | 276 | 824
Not Completed | 54 | 161
Not completed — Protocol Violation | 6 | 18
Not completed — Adverse Event | 10 | 46
Not completed — Lack of Efficacy | 1 | 2
Not completed — Withdrawal by Subject | 15 | 36
Not completed — Lost to Follow-up | 13 | 39
Not completed — Death | 2 | 2
Not completed — Decision by the Sponsor | 4 | 8
Not completed — Other than specified above | 3 | 10

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Placebo: Two subcutaneous injections of Placebo (for Rilonacept) as a loading dose on Day 1 followed by a single injection qw from Week 1 to Week 15.
- Total: Total of all reporting groups
Arm/Group | Placebo | Rilonacept 160 mg | Total
Number analyzed (Participants) | 330 | 985 | 1315
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (10.55) | 52.8 (11.48) | 52.7 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 128 | 161
  Male | 297 | 857 | 1154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 38 | 49
  Not Hispanic or Latino | 319 | 947 | 1266
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 7 | 9
  Asian | 47 | 115 | 162
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 70 | 202 | 272
  White | 210 | 658 | 868
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence in a participant who received investigational medicinal product (IMP) was considered an AE without regard to possibility of causal relationship with this treatment. Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during on-treatment period (time from the administration of first dose of study drug up to 35 days after the last dose of study drug). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Baseline up to Week 20
Population: Safety analysis set that included all participants who received any study drug and safety analyses were based on the treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 330 | 985
percentage of participants
  With at least 1 TEAE | 59.1 | 66.6
  With TEAEs related to study drug | 13.0 | 27.5
  With serious TEAEs | 3.9 | 3.1
  With TEAEs resulting in drug withdrawal | 3.3 | 5.0
  With serious TEAEs resulting in drug withdrawal | 1.8 | 1.1
  With TEAEs leading to study discontinuation | 3.0 | 4.7
  With serious TEAE leading to study discontinuation | 1.5 | 1.0
  Treatment emergent deaths | 0.3 | 0.2

2. Secondary Outcome: Number of Gout Flares Per Participant Assessed From Day 1 to Day 112 (Week 16)
Description: A gout flare was defined as participant reported acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Number of gout flares per participant was reported for this outcome measure. For drop-outs, only flares occurred before Day 112 were counted, regardless whether the flares occurred during the treatment period or not.
Time Frame: Day 1 to Day 112 (Week 16)
Population: Full analysis set (FAS) that included all randomized participants who received any study medication, and was based on the treatment allocated by the Interactive voice response system (IVRS) at randomization (as randomized). Here, number of participants analyzed=participants with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: Gout flares
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 323 | 952
Gout flares | 1.73 (2.69) | 0.51 (1.17)

3. Secondary Outcome: Percentage of Participants With at Least One Flare From Day 1 to Day 112 (Week 16)
Description: A gout flare was defined as participant reported acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Percentage of participants with at least one gout flare was reported for this outcome measure. For drop-outs, only flares occurred before Day 112 were counted, regardless whether the flares occurred during the treatment period or not.
Time Frame: Day 1 to Day 112 (Week 16)
Population: FAS that included all randomized participants who received any study medication, and was based on the treatment allocated by the IVRS at randomization (as randomized).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 330 | 985
percentage of participants | 51.1 | 25.7

4. Secondary Outcome: Percentage of Participants With at Least Two Flares From Day 1 to Day 112 (Week 16)
Description: A gout flare was defined as participant reported acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Percentage of participants with at least two gout flare was reported for this outcome measure. For drop-outs, only flares occurred before Day 112 were counted, regardless whether the flares occurred during the treatment period or not.
Time Frame: Day 1 to Day 112 (Week 16)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 330 | 985
percentage of participants | 34.7 | 11.7

5. Secondary Outcome: Number of Gout Flare Days Per Participant From Day 1 to Day 112 (Week 16)
Description: A gout flare was defined as participant reported acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Number of gout flares per participant was reported for this outcome measure. Flare days were counted up to Week 16, regardless of whether or not the flares occurred during the treatment period.
Time Frame: Day 1 to Day 112 (Week 16)
Population: FAS that included all randomized participants who received any study medication, and was based on the treatment allocated by the IVRS at randomization (as randomized). Here, number of participants analyzed=participants with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: Gout flare Days
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 323 | 952
Gout flare Days | 7.66 (11.79) | 2.66 (7.69)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 20) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from the administration of first dose of study drug up to 35 days after the last dose of study drug).
Arm/Group | Placebo | Rilonacept 160 mg
Serious Adverse Events (participants affected / at risk) | 13/330 | 31/985
Other Adverse Events (participants affected / at risk) | 74/330 | 266/985
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=330) | Rilonacept 160 mg (N=985)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=330) | Rilonacept 160 mg (N=985)
Injection site erythema (General disorders) | 1 (1) | 61 (195)
Accidental overdose (Injury, poisoning and procedural complications) | 20 (21) | 54 (61)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (41) | 65 (85)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (21) | 52 (74)
Headache (Nervous system disorders) | 26 (45) | 90 (169)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI/Institution will provide a copy of any publication to Sponsor prior to submission for review. Sponsor may request to remove confidential information from submission, provided that removal does not preclude the complete and accurate presentation and interpretation of the study results.